CLINICAL TRIAL: NCT02442193
Title: Individual Placement and Support (IPS) for Patients With Offending Histories: Feasibility of an Evidence-based Approach in Forensic Mental Health Settings
Brief Title: Individual Placement and Support for Patients With Offending Histories
Acronym: IPSOH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by the funder due to low recruitment rates.
Sponsor: Nottinghamshire Healthcare NHS Trust (Other Government)
Collaborators: University of Nottingham (Other); University of Southampton (Other); University of Leicester (Other); Institute of Mental Health Nottingham (Other)
Responsible Party: Principal Investigator, Najat Khalifa, Associate Professor, Nottinghamshire Healthcare NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KHALIFA/020415; PB-PG-1013-32093 (Other Grant/Funding Number: NIHR - Research for Patient Benefit (RfPB))
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Employment, Supported; Treatment as Usual
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Placement and Support (Experimental): Individual Placement and Support
  Interventions: Other: Individual Placement and Support
- Treatment as Usual (No Intervention): Treatment as Usual is comprised of routine clinical care.

INTERVENTIONS:
Other: Individual Placement and Support — Individual Placement and Support is a form of supported employment.
  Arms: Individual Placement and Support

SUMMARY:
The overall aim of the study is to assess the feasibility of conducting a Randomized Controlled Trial (RCT) to evaluate the effectiveness of Individual Placement and Support (IPS) in improving employment rates and associated psychosocial outcomes in forensic psychiatric populations.

DETAILED DESCRIPTION:
This is a feasibility trial which aims to assess the feasibility of conducting a full Randomized Controlled Trial (RCT) to evaluate the effectiveness of Individual Placement and Support (IPS) in improving employment rates and associated psychosocial outcomes in forensic psychiatric populations.

Given that IPS is a complex intervention, the design of this study has drawn from the principles set out in the UK Medical Research Council (MRC) Guidance on developing and evaluating complex interventions by defining three major research strands in order to achieve the specific objectives of the study as follows:

A. Implementation of IPS in community forensic services: The specific objective of this strand is to embed the IPS model in the community forensic services in which the feasibility study will be carried out (aided by an IPS Expert), by bringing an employment specialist into clinical teams, raising awareness about IPS within the organization, forming links with IPS services in the area and developing links with employers, as well as conducting IPS fidelity reviews.

B. Feasibility Cluster Randomized Controlled Trial (RCT): The specific objectives of this strand are to estimate the parameters required to design a full RCT including:

1. Means and standard deviations of the key outcome measures in order to benchmark potential effect sizes and enable sample size calculations.
2. The feasibility of randomization, recruitment and retention rates to the IPS and controls;
3. The suitability of the key outcome measures with respect to: reliability, acceptability, and distribution of the scores.

C. Process Evaluation: This will be carried out in parallel with the other two strands to meet other specific objectives by using the following methods:

1. Qualitative interviews with staff to identify the structural, legal, organizational and individual-level to barriers and facilitators to implementation of IPS in community forensic services.
2. Fidelity Reviews to assess the extent to which the services follow the principles of IPS and to assess how well the employment specialist functions within the community forensic services.
3. Qualitative interviews with patients assigned to IPS in order to assess their general views of IPS, benefits from participating, disadvantages from or dislikes about participating and barriers and facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years
* Patients (females and males) on the caseload of the community forensic services

Exclusion Criteria:

* Patients unable to provide informed consent
* Patients not eligible to work in the UK
* Patients currently in open employment
* Patients who do not wish to work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Open Employment: Proportion of people in open employment | 12 Months
  Proportion of people in open employment at 12 month follow-up

SECONDARY OUTCOMES:
Number of hours worked | 12 Months
  Number of hours worked at 12 month follow-up
Mental health as measured using the Brief Psychiatric Rating Scale (BPRS) | Baseline, 6 and 12 Months
  Measured using the Brief Psychiatric Rating Scale (BPRS)
Social Functioning as measured using the Social Functioning Questionnaire (SFQ) | Baseline, 6 and 12 Months
  Measured using the Social Functioning Questionnaire (SFQ)
Self-Esteem as measured using the Rosenberg's Self Esteem Scale | Baseline, 6 and 12 Months
  Measured using the Rosenberg's Self Esteem Scale
Work Limitations as measured using the Work Limitation Questionnaire | Baseline, 6 and 12 Months
  Measured using the Work Limitation Questionnaire
Quality of life as measured using SF-12v2 | Baseline, 6 and 12 Months
  Health-related quality of life as measured using SF-12v2
Economic Costing as measured using the Client Service Receipt Inventory (CSRI) | Baseline, 6 and 12 Months
  Measured using the Client Service Receipt Inventory (CSRI)
Re-offending rates | Baseline and 18 Months
  Re-offending rates
Number of days in open employment | 12 months
  Number of days in open employment at 12 months
Quality of life as measured using the EQ5-D | Baseline, 6 and 12 months
  Health-related quality of life as measured using the EQ5-D

CONTACTS AND LOCATIONS:
Overall Officials: Najat R Khalifa, DM, Principal Investigator — Nottinghamshire Healthcare NHS Trust
Locations (1):
- Nottinghamshire NHS Foundation Trust, Nottingham, United Kingdom

REFERENCES:
- [Result] Khalifa N, Talbot E, Schneider J, Walker DM, Bates P, Bird Y, Davies D, Brookes C, Hall J, Vollm B. Individual placement and support (IPS) for patients with offending histories: the IPSOH feasibility cluster randomised trial protocol. BMJ Open. 2016 Jul 22;6(7):e012710. doi: 10.1136/bmjopen-2016-012710. PMID 27449894
- [Derived] Khalifa N, Talbot E, Barber S, Schneider J, Bird Y, Attfield J, Bates P, Walker DM, Vollm B. A Feasibility Cluster Randomized Controlled Trial of Individual Placement and Support (IPS) for Patients With Offending Histories. Front Psychiatry. 2020 Jan 13;10:952. doi: 10.3389/fpsyt.2019.00952. eCollection 2019. PMID 31998164
- See also: Study Protocol — http://bmjopen.bmj.com/content/6/7/e012710